CLINICAL TRIAL: NCT04857164
Title: A Prospective Study of Pembrolizumab Combined with Chemotherapy (cisplatin or Carboplatin + Albumin-bound Paclitaxel) in First-line Therapy for Patients with Recurrent and Metastatic Squamous Cell Carcinoma of the Head and Neck
Brief Title: Study of Pembrolizumab Combined with Chemotherapy in the First Line Therapy for R/M HNSCC in China
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yuankai Shi (Other)
Responsible Party: Sponsor-Investigator, Yuankai Shi, Director, Head of Oncology, Chief physician, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Organization: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KTP-001
Record Dates: First submitted 2021-04-14; First posted 2021-04-23 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: Head and Neck Cancer; immune therapy; Pembrolizumab combined with chemotherapy
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms | interventions — Drug Therapy; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pembrolizumab combined with Chemotherapy (Experimental): Chemotherapy regimen* is as follows, selected by the investigator, 3 weeks (21 days) is a cycle，combined with pembrolizumab 200 mg intravenously on day 1, every 21 days is a treatment cycle until the disease progresses or the toxicity cannot be tolerated(Less than or equal to 35 cycle)
  *1) Cisplatin(75 mg/m2) + albumin-bound paclitaxel(260 mg/m2) 2)Cisplatin(25 mg/m2,d1-d3) + albumin-bound paclitaxel(260 mg/m2) 3)Carboplatin(AUC5) + Albumin-bound Paclitaxel(260 mg/m2)
  Interventions: Drug: Pembrolizumab combined with Chemotherapy

INTERVENTIONS:
Drug: Pembrolizumab combined with Chemotherapy — Pembrolizumab (formerly lambrolizumab, brand name Keytruda) is a humanized antibody used in cancer Chemotherapy regimen is selected by the investigator immunotherapy. This includes to treat melanoma, lung cancer, head and neck cancer, Hodgkin lymphoma, and stomach cancer.
  Other Names: keytruda and Chemotherapy

SUMMARY:
This trial is main evaluate the efficacy and safety of pembrolizumab combined with chemotherapy in the first-line treatment of Chinese patients with recurrent or metastatic head and neck squamous cell carcinoma

DETAILED DESCRIPTION:
This trial is a single-center, prospective phase II clinical study, which mainly evaluates the efficacy and safety of first-line treatment with pembrolizumab combined with chemotherapy in patients with recurrent and/or metastatic head and neck squamous cell carcinoma

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign written informed consent before screening;
2. Age 18~75 years old;
3. ECOG physical status score 0-1 points;
4. Head squamous cell carcinoma (HNSCC) diagnosed by histology or cytology, the primary site is oral cavity, oral cavity Throat, lower throat or throat;
5. Recurrent and/or metastatic HNSCC without indications for local radical treatment;
6. According to the evaluation criteria for the efficacy of solid tumors (RECIST version 1.1), there is at least one measurable lesion, right For lesions that have received radiotherapy in the past, only if there is clear disease progression 3 months after the end of radiotherapy, can it be Was selected as the target lesion;
7. There are a large number of tumor tissue samples for PD-L1 immunohistochemical detection;
8. The expected survival period exceeds 3 months;
9. The main organs function normally, that is, they meet the following standards:

   I. Blood routine (not receiving blood transfusion 14 months before screening examination, erythropoietin (EPO), granulocyte set Fall stimulating factor (G-CSF) or granulocyte-macrophage colony stimulating factor (GM-CSF) treatment): neutral Granulocyte ≥1.5×l09
   * L, platelets ≥100×109
   * L, hemoglobin≥90g/L; ii. Liver function: alanine aminotransferase (ALT) and aspartate aminotransferase (AST), ALT and AST ≤ 3 for those without liver metastasis ×ULN, ALT and AST for liver metastases≤5×ULN; total bilirubin (TBIL)≤1.5×ULN (Gilbert Syndrome patients, ≤3×ULN); iii. Renal function: Serum creatinine (Cr)≤1.5×ULN or tendon clearance (Ccr)≥50ml/min (connect Residues treated with carboplatin) or ≥60ml/min (residuals treated with cisplatin); iv. Coagulation function: activated partial thromboplastin time (APTT), international normalized ratio (INR), thrombin Original time (PT)≤1.5×ULN; v. Heart echocardiogram: left ventricular ejection fraction (LVEF) ≥50%;
10. Women should agree to use contraceptive measures (such as intrauterine birth control) during the study period and within 6 months after the study ends.

Device [IUD], contraceptive pill or condom); 7 diabetes blood pregnancy test was negative before study enrollment, and it must be non-Breastfeeding patients; males should agree to use contraceptive measures during the study period and within 6 months after the end of the study period patient.

Exclusion Criteria:

1. Patients who are suitable for local treatment and are willing to local treatment;
2. Have received systemic chemotherapy, but does not include treatment for locally advanced disease as a part of multimodal treatment Chemotherapy (the end of this treatment must be more than 6 months after the first trial medication); Note: Multimodal therapy includes induction chemotherapy, concurrent radiotherapy and chemotherapy and adjuvant chemotherapy.
3. Locally advanced head and neck squamous cell carcinoma multimodal treatment is completed within 6 months of disease progression;
4. Have received anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137 or anti-CTLA-4 antibodies or targeting effects in the past Any other antibody or drug immunotherapy in T cell co-stimulation or immune checkpoint pathway;
5. Other malignant tumors have occurred within 5 years or at the same time during the current period, except for cured cervical carcinoma in situ, non- Skin cancer of melanoma or other tumors/cancers that have undergone radical treatment and have no signs of disease for at least 5 years;
6. Received cetuximab treatment within 6 months before the first administration;
7. According to the standard of common adverse event term (NCI CTCAEv5.0), peripheral neuropathy has been ≥2 grade;
8. With known active central nervous system metastasis (CNS) and/or cancerous meningitis: previous treatment Subjects with brain metastases treated for treatment can participate in the study, provided that they are clinically stable for at least 2 weeks and there are no new or enlarged brains.

   Evidence was transferred, and steroids were discontinued 14 days before study drug administration. The stable brain metastasis in this definition should be in Determine before the first administration of the study drug. Subjects with asymptomatic brain metastases (ie no neurological symptoms, no need Corticosteroids, and no lesions> 1.5cm) can participate, but the brain needs to be regularly performed as a disease site Film degree exam;
9. Did not recover from any acute effects of previous surgery, chemotherapy or radiotherapy, that is, did not fall to ≤1 grade (NCI CTCAEv5.0) subjects (except for hair loss). If the nutritional status is stable, allow previous radiotherapy and/or surgery Chronic late toxicity (pharyngeal/larynx toxicity, ie dry mouth, abnormal speech, swallowing, etc.);
10. Any component of the studied drug or preparation has caused severe allergic reactions, including known Severe allergic reaction to Longan antibody (NCI CTCAEv5.0≥3);
11. Have received anti-tumor drug treatment (such as chemotherapy, hormone therapy, immune Disease treatment, antibody treatment, radiotherapy, etc.), except for palliative radiotherapy for bones to relieve pain;
12. Chinese herbal medicine or Chinese patent medicine receiving anti-tumor treatment ≤1 week before the first administration;
13. Have received major surgery within 4 weeks before the first administration or are expected to undergo major surgery during the study period;
14. Immunosuppressive drugs need to be used 2 weeks before the first administration or within 2 weeks or during the study period. The following conditions are excluded:

    1. Intranasal, inhaled, topical steroid or topical steroid injection (such as intra-articular injection);
    2. Physiological dose of systemic corticosteroids (≤10mg/day prednisone or equivalent dose);
    3. Short-term (≤7 days) use of steroids to prevent or treat non-autoimmune allergic diseases;
15. Subjects who are known to have active or have a history of autoimmune diseases that are likely to relapse (such as:

    Systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, autoimmune thyroid disease, multiple Sexual sclerosis, vasculitis, glomerulitis, etc.), or high risk (such as receiving an organ transplant and requiring immunotherapy) Of patients. However, the following patients are allowed to join the group: patients with type I diabetes who are in stable condition after using a fixed dose of insulin Those; autoimmune hypothyroidism requiring only hormone replacement therapy; no need for systemic therapy Skin diseases (such as eczema, skin rashes that account for less than 10% of the body surface, psoriasis without ophthalmological symptoms, etc.);
16. Subjects with known history of interstitial lung disease, history of non-infectious pneumonia, or high suspicion of interstitial lung disease Those who have previously had drug-induced or radiation non-infectious pneumonia but asymptomatic subjects are allowed to enter the group;
17. A history of human immunodeficiency virus infection (positive HIV test), or other acquired or congenital Immunodeficiency disease, or history of organ transplantation, or history of stem cell transplantation;
18. The hepatitis B or C virological examination at the time of screening meets any of the following:

    1. HBsAg positive, and peripheral blood hepatitis B virus deoxyribonucleic acid (HBV DNA) titer ≥104 Copy number/ml or ≥2000 IU/ml;
    2. HCV antibody is positive, and HCV-RNA is higher than the detection limit of the analysis method;
19. Within 2 weeks or 2 weeks before the first administration, the subject has an active infection that requires systemic treatment or is uncontrollable Infection (except for simple urinary tract infection or upper respiratory tract infection);
20. Live virus vaccine was vaccinated within 4 weeks before the first dose. Allows vaccination against seasonal influenza that does not contain live viruses seedling;
21. Serous effusions (such as pleural effusions and pleural effusions) with clinical symptoms that require clinical intervention or stable time less than 4 weeks ascites);
22. Known to be accompanied by serious medical diseases, such as heart function abnormalities of grade III and above (New York Heart Association [NYHA]), cardiovascular diseases such as ischemic heart disease (such as myocardial infarction or angina pectoris), or before the first administration 3 A history of myocardial infarction within months, and poorly controlled diabetes (fasting blood glucose ≥ 10mmol/L) or poorly controlled hypertension (systolic blood pressure ≥160mmHg and/or diastolic blood pressure ≥100mmHg);
23. Medical or psychiatric history or laboratory abnormal history that may interfere with the interpretation of results;
24. The subject is currently enrolled in other research equipment or research drug research, or is away from other research drugs Or the study device is out of use for less than or equal to 4 weeks;
25. The subject is known to be addicted to alcohol or drugs;
26. The researcher believes that the subjects have other conditions that may affect their compliance with the protocol and the evaluation of research indicators.

Circumstances, subjects who are not suitable to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-04-30 (Actual); Primary Completion 2023-08-20 (Actual); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
objective response rate(ORR) | 18 weeks
  To evaluate the objective response rate of pembrolizumab combined with chemotherapy in the first-line treatment of Chinese patients with recurrent and or metastatic head and neck squamous cell carcinoma

SECONDARY OUTCOMES:
progression free survival(PFS) | 4 year
  To evaluate the progression free survival (PFS) of pembrolizumab combined with chemotherapy in the first-line treatment of Chinese patients with recurrent and or metastatic head and neck squamous cell carcinoma
disease control rate (DCR) | 4 year
  To evaluate the disease control rate of pembrolizumab combined with chemotherapy in the first-line treatment of Chinese patients with recurrent and or metastatic head and neck squamous cell carcinoma
duration of response (DOR) | 4 year
  To evaluate the duration of response (DOR) of pembrolizumab combined with chemotherapy in the first-line treatment of Chinese patients with recurrent and or metastatic head and neck squamous cell carcinoma
progression free survival rate(PFS rate) | 6 months and 12 months
  PFS rates at 6 and 12 months
overall survival (OS) | 4 year
  To evaluate the survival time (OS) of pembrolizumab combined with chemotherapy in the first-line treatment of Chinese patients with recurrent and or metastatic head and neck squamous cell carcinoma

OTHER OUTCOMES:
Tumor related biomarkers | 4 year
  Biomarker analysis related to blood or tumor tissue before and after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, MD, Principal Investigator — Cancer Institute/Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College
Locations (1):
- National Cancer Center/Cancer Hospitial,Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No